CLINICAL TRIAL: NCT03673527
Title: Open-label, Non-randomised, Single-centre, Multiple-dose, Phase 1, Pharmacokinetic Trial With a Topical Formulation of Tacrolimus in Healthy Subjects
Brief Title: Tacrolimus Blood Levels After Topical Application of Tacrolimus on Healthy Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LP0121-1388; 2018-001959-12 (EudraCT Number)
Record Dates: First submitted 2018-08-07; First posted 2018-09-17 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: open-label; multiple-dose; non-randomised; non-comparative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- topical formulation of tacrolimus (Experimental)
  Interventions: Drug: topical formulation of tacrolimus

INTERVENTIONS:
Drug: topical formulation of tacrolimus — Topical application of tacrolimus twice daily for 14 days (one dose on Day 14).

SUMMARY:
This is a phase I trial to evaluate tacrolimus blood levels after topical application of tacrolimus twice daily on healthy skin.

DETAILED DESCRIPTION:
The purpose of this trial is to assess the safety of a topical formulation of tacrolimus.

Tacrolimus is commonly used in T-cell medicated diseases. It is expected that 24 subjects will be enrolled in the trial and will be assigned to receive topical application of tacrolimus twice daily for 14 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female subjects between 18 and 60 years of age, with a body mass index (BMI) between 18.5 and 30 kg/m2 inclusive
* Female subjects of childbearing potential must be confirmed not pregnant at the screening visit and use highly effective contraception during the trial.

Key Exclusion Criteria:

* Treatment with the following medications: Topical immunosuppressive drugs (e.g. tacrolimus, corticosteroids), systemic immunosuppressive/immunomodulating drugs
* Extensive UV radiation or sunlight on the application sites
* Skin diseases
* Wounded or damaged skin at the application site
* Immunosuppressed or immunocompromised individuals
* Renal or hepatic impairment or insufficiency
* Known allergy or known or suspected hypersensitivity to any component(s) of the topical formulation of tacrolimus
* Female subjects who are pregnant or lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Twelve Hours (AUC0-12) of tacrolimus on Days 1 and 14 | Up to Day 14
Maximum Observed Drug Concentration (Cmax) of tacrolimus | On Days 1 and 14

SECONDARY OUTCOMES:
Number of adverse events (AEs) up to Day 21 | Day -22 to Day 21
Number of subjects with AEs up to Day 21 | Day -22 to Day 21
Absolute values of systolic and diastolic blood pressure at Days 1, 2, 14, and 21 summarised by mean and standard deviation | Day 1 to Day 21
  Measurement unit: mmHg
Absolute values of pulse at Days 1, 2, 14, and 21 summarised by mean and standard deviation | Day 1 to Day 21
  Measurement unit: bpm
Absolute values of body temperature at Days 1, 2, 14, and 21 summarised by mean and standard deviation | Day 1 to Day 21
  Measurement unit: °C
Changes in systolic and diastolic blood pressure from baseline to Day 21 summarised by mean and standard deviation | Day 1 to Day 21
  Measurement unit: mmHg
Changes in pulse from baseline to Day 21 summarised by mean and standard deviation | Day 1 to Day 21
  Measurement unit: bpm
Changes in body temperature from baseline to Day 21 summarised by mean and standard deviation | Day 1 to Day 21
  Measurement unit: °C
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of tacrolimus on Day 14 | Day 1 to Day 14
Apparent Terminal Half-life (t1/2) of tacrolimus on Day 14 | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Investigational site, Neu-Ulm, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No